CLINICAL TRIAL: NCT03798106
Title: A Phase II Trial of Pazopanib and Durvalumab for Metastatic Soft Tissue Sarcoma
Brief Title: A Study of Pazopanib and Durvalumab for Metastatic Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Principal Investigator, Hyo Song Kim, professor, Yonsei University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2018-0743
Record Dates: First submitted 2019-01-07; First posted 2019-01-09 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — durvalumab; pazopanib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- durvalumab+pazopanib (Experimental): Durvalumab 1500mg IV 1hr q3weeks Pazopanib 800mg QD PO q3wwks
  Interventions: Drug: Durvalumab, pazopanib

INTERVENTIONS:
Drug: Durvalumab, pazopanib — Durvalumab 1500mg IV 1hr q3weeks Pazopanib 800mg QD PO q3wwks

SUMMARY:
Pazopanib is an angiogenesis inhibitor targeting VEGFR-1, -2, and -3; PDGFR-α and -β; and the receptor c-Kit, and is indicated for the treatment of subjects with advanced renal cell carcinoma (RCC) and advanced STS. For this orphan tumor, STS, PD-L1 targeting may be a promising strategy and favorable toxicity may warrant further combination.

DETAILED DESCRIPTION:
Pazopanib is an angiogenesis inhibitor targeting VEGFR-1, -2, and -3; PDGFR-α and -β; and the receptor c-Kit, and is indicated for the treatment of subjects with advanced renal cell carcinoma (RCC) and advanced STS. Pro-angiogenic factors suppress various immune functions whereas antiangiogenic agents have potential to modulate the tumor microenvironment and improve immunotherapy. An analysis of patients with RCC treated with pazopanib demonstrated that elevated expression of PD-L1 correlates with shorter PFS. Investigator also identified 43% of PD-L1 expression in STS and PD-L1 expression had worse overall survival (5-year survival rate: 48% in PD-L1 positive vs. 68% in PD-L1 negative, p=0.015). In detail, PD-L1 expression was reported 52.6% in synovial sarcoma, 37.6% in rhabdomyosarcoma, and 100% in epithelioid sarcoma. For this orphan tumor, STS, PD-L1 targeting may be a promising strategy and favorable toxicity may warrant further combination.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed STS progression to 1 or 2 prior chemotherapy
2. Age > 18 years at time of study entry.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
4. Measurable disease by Response Evaluation Criteria in Solid Tumors Version 1.1
5. Body weight >30kg
6. Adequate laboratory findings
7. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients.
8. Patient is willing and able to comply with the protocol for the duration of the study
9. Must have a life expectancy of at least 12 weeks
10. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
11. Patients with evidence of portal hypertension (including splenomegaly detected radiographically) or any prior history of variceal bleeding must have had endoscopic evaluation within the 3 months immediately prior to enrollment, and the findings do not represent a high bleeding risk.

Exclusion Criteria:

1. More than 4 prior cytotoxic regimens
2. Participation in another clinical study with an investigational product during the last 2 weeks
3. Receipt of the last dose of anticancer therapy 14 days prior to the first dose of study drug
4. Any previous treatment with a PD1 or PD-L1 inhibitor (including durvalumab) and/or pazopanib
5. Mean QT interval corrected for heart rate (QTc) >480 ms calculated from 3 electrocardiograms (ECGs) using Fridericia's Correction
6. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria
7. Any concurrent chemotherapy, biologic, or hormonal therapy for cancer treatment within 2 weeks prior to entering the study. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable
8. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug
9. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP.
10. History of allogenic organ transplantation.
11. Active or prior documented autoimmune or inflammatory disorders
12. Uncontrolled intercurrent illness
13. History of active infection
14. History of another primary malignancy
15. History of leptomeningeal carcinomatosis who are neurologically unstable or have required active treatment
16. Receipt of live attenuated vaccine within 30 days prior to the first dose of investigational product(IP).
17. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose.
18. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
19. No history of any of the following in the past 6 months: cardiac angioplasty or stenting, myocardial infarction, unstable angina, coronary artery bypass graft surgery, symptomatic peripheral vascular disease class III or IV congestive heart failure, as defined by the New York Heart Association), thromboembolic events

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate | 12 weeks
  antitumor efficacy of durvalumab and pazopanib

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No